CLINICAL TRIAL: NCT03310736
Title: Evaluation of the Intrinsic Hepcidin IDx™ Test to Detect Iron Deficiency and Predict Response to Oral Iron Therapy in Adolescents and Young Adults
Brief Title: Serum Hepcidin Immunoassay - Laboratory to Marketplace
Status: Completed | Type: Observational
Sponsor: Intrinsic LifeSciences, LLC (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ILS-0001
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Anemia, Iron Deficiency
Keywords: iron deficiency; anemia; hepcidin
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Any remaining blood, serum or plasma specimens will be stored in a deidentified fashion in an annotated repository at IntrinsicDX for future research on ID and anemia to be conducted by the participating investigators. The key to the deidentified specimens will be held at BCH and will not be shared with the sponsor. After the primary study has been published, the data will be anonymized by destroying any deidentifier keys.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intrinsic Hepcidin IDx™ Test — ILS scientists developed the bioanalytical method for quantitation of human serum hepcidin using a Beckman FX automated liquid handling platform. The method uses a competitive ELISA format that has a proprietary sensitive and specific monoclonal antibody to hepcidin that captures native hepcidin in a sample. During the reaction a competition between a synthetic, bioactive, biotinylated hepcidin tracer and native hepcidin occurs. Bound biotinylated tracer is detected with a streptavidin-HRP conjugate and TMB substrate. Quantitation is based on an eight-point standard curve using validated, synthetic hepcidin calibrators. The standard curve and the hepcidin concentrations of patients samples are calculated using 4-parameter logistic curve fitting (Prism; Graphpad, Inc., La Jolla, CA). Serum hepcidin concentrations are expressed in ng/ml serum.

SUMMARY:
This is a single center, prospective, observational study to demonstrate the clinical validity of the Intrinsic LifeSciences (ILS) Intrinsic Hepcidin IDx™ Test in the diagnosis and management of iron deficiency (ID) in adolescents and young adults. This test is considered non-significant risk.

DETAILED DESCRIPTION:
This observational study is composed of two phases, and no investigational intervention agent. Oral iron therapy will be recommended by each subject's primary care clinician or his/her designate according to standard clinical care. There is no randomization. Subjects will be screened for enrollment by study personnel.

Diagnostic Testing Phase (Study Visit 1). Enrolled subjects will have a study blood draw. Enrolled subjects will be assessed for presence of ID as defined by the reference standard: ID: Ferritin < 20 ng/mL.

Enrolled subjects will be assessed for presence of anemia as defined by: Anemia - Hemoglobin ≤ 11 g/dL

Those determined to have ID and/or anemia and are prescribed oral iron therapy by their clinician will continue to the next phase in the study. For those without ID or anemia, or who meet Observation of Treatment Phase exclusion criteria, study participation will be complete. The expected duration of subject involvement for the Diagnostic Testing Phase is 1 week.

Observation of Treatment Phase (Study Visits 2 and 3). Subjects identified as having ID and/or anemia and who have been prescribed oral iron therapy by their physician according to standard of care, and do not meet Observation of Treatment Phase exclusion criteria, will continue to the Observation of Treatment Phase of the study.

The optimal dose, frequency, and timing of oral iron therapy are unknown and are based more on clinical experience than evidence. In 1998, based on expert opinion, the Centers for Disease Control (CDC) suggested 3 mg/kg/day of elemental iron for treatment of IDA in children. Patients with ID who do not have anemia (LID) should also have their iron stores repleted with treatment dose iron supplement. Given the effects of acute/chronic disease on serum ferritin and the dietary/diurnal variation of serum iron/TfSat, the absence of biochemical evidence of ID on a single measure does not rule out ID that may respond to empiric supplementation. Therefore, patients with anemia but without biochemical evidence of ID (AneID) may have masked ID and treatment with a finite course of supplemental iron therapy is unlikely to result in harm and may improve hemoglobin. Thus, we expect all subjects with ID and/or anemia will be recommended treatment by their clinician with ferrous sulfate at treatment at standard doses for adolescents and young adults of 3-5 mg elemental iron/kg/day, up to a maximum of 195 mg of elemental iron per day.

Investigators will provide responsible clinicians with recommendations for ferrous sulfate treatment along with references to relevant clinical guidelines and research. The clinicians will be asked to provide the research team confirmation that the patient followed the oral iron treatment recommendations. If they did not, they will be asked to indicate what treatment, if any, they did advise for the subject.

Subjects who continue to the Observation of Treatment Phase will have two follow-up visits and laboratory testing, including a study draw for hepcidin at each visit, to assess response to oral iron supplementation at:

* 4-5 weeks (+/- 7 days) of therapy, and
* 12 weeks (+/- 7 days) of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 11 years
* Subjects must give informed assent/ consent prior to the blood draw. Subjects that are minors (<18 years) must have a parent or guardian give informed consent and the subject must give assent to participate in the study.
* Willing to comply with all oral iron supplementation and follow up visits if they move to the Observation of Treatment Phase.
* Able to communicate in English.

Exclusion Criteria:

* Acute febrile illness (Temp ≥100.4°F (38°C), or acute otitis media, gastroenteritis, pharyngitis or other URI, within the previous one week.
* History of known hemoglobinopathy (e.g., thalassemia trait or sickle cell)
* Any parenteral iron received in the 30 days prior to enrollment.
* Presently taking oral iron supplements (except for iron as part of multivitamin or oral contraceptive pill) or has taken it in the 30 days prior to enrollment.
* An allergy or hypersensitivity to oral iron sulfate.
* Has received a blood transfusion in the 90 days prior to enrollment.
* Any investigational drug use in the 30 days prior to enrollment.
* Any known malignancy.
* Receiving dialysis.
* Known to be pregnant or currently breast-feeding.
* Any lab abnormality, medical condition, or psychiatric disorder which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The primary care clinic at Boston Children's Hospital (BCH) Adolescent/Young Adult (AYA) Clinic, BCH Sports Medicine Clinic, or at Boston Children's Physicians Weymouth
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the Intrinsic Hepcidin IDx test | 12 weeks
  To demonstrate the diagnostic accuracy of the Intrinsic Hepcidin IDx TestTM to diagnose ID in adolescents and young adults, where diagnostic accuracy is defined by the lower 95% confidence interval on sensitivity (Se) being not less than 70% and the lower 95% confidence interval on specificity (Sp) not being less than 70%.

SECONDARY OUTCOMES:
Prediction of Response to Oral Iron Therapy | 12 weeks
  To evaluate the ability of the Intrinsic Hepcidin IDx TestTM to predict a response to oral iron therapy in adolescents and young adults with ID
Predict Therapeutic Response to Oral Iron Therapy | 12 weeks
  To evaluate the ability of the Intrinsic Hepcidin IDx TestTM to predict a therapeutic response to oral iron therapy in adolescents and young adults with anemia and no biochemical evidence of iron deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Heeney, MD, Principal Investigator — Physician; Lydia A Shrier, MD, MPH, Principal Investigator — Physician
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No